CLINICAL TRIAL: NCT02741206
Title: Bellevue ROSE: Preventing Postpartum Depression in Prenatal Care
Brief Title: Preventing Postpartum Depression in Prenatal Care
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 15-01130
Record Dates: First submitted 2016-03-30; First posted 2016-04-18 (Estimated); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Post-partum Depression
Keywords: psycho-education; maternal depression; Reach Out Stay Strong Essentials
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- High Risk PTSD Group 1 (Active Comparator): Forty women who are eligible for the study will be randomized into either the Bellevue ROSE intervention (treatment group) or a psycho-education session and usual, standard of care (control group 1)
  Interventions: Behavioral: Bellevue ROSE Intervention; Behavioral: Psycho-education session and usual, Standard of care Control
- High Risk PTSD Group 2 (Active Comparator): Forty women who are eligible for the study will be randomized into either the Bellevue ROSE intervention (treatment group) or a psycho-education session and usual, standard of care (control group 1)
  Interventions: Behavioral: Bellevue ROSE Intervention; Behavioral: Psycho-education session and usual, Standard of care Control
- Low Risk PTSD Control (Experimental): Twenty additional women, who are at lower risk and thus not eligible for randomization, will also receive one psycho-education session and usual care (control group 2).
  Interventions: Behavioral: One Psycho-education session and usual, standard of care Control

INTERVENTIONS:
Behavioral: Bellevue ROSE Intervention
  Arms: High Risk PTSD Group 1; High Risk PTSD Group 2
Behavioral: Psycho-education session and usual, Standard of care Control — Psycho Education and usual, standard of care
  Arms: High Risk PTSD Group 1; High Risk PTSD Group 2
Behavioral: One Psycho-education session and usual, standard of care Control
  Arms: Low Risk PTSD Control

SUMMARY:
This is randomized control trial of a brief intervention called Bellevue ROSE (Reach Out Stay Strong Essentials). Bellevue ROSE is a manualized and highly structured interpersonal intervention that provides women with psycho-education about maternal depression and strategies for strengthening social support and connectedness. Investigators use motivational interviewing strategies to improve treatment compliance and resource acquisition

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Women who score between 5-19 on the PHQ-9 and >23 on the ANRQ

Exclusion Criteria:

* Women who score <5 or >19 on the PHQ-9
* Women who are currently suicidal, active substance users, currently experiencing domestic violence, or have a current or past history of bipolar or psychotic disorder diagnosis.
* Women who are currently in treatment for psychotherapy.
* Unable to speak and/or understand English proficiently
* Unable to provide informed consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06; Primary Completion 2017-07-20 (Actual); Study Completion 2017-07-20 (Actual)

PRIMARY OUTCOMES:
Depression severity measured by Patient Health Questionnaire (PHQ-9) | 6 Months
Measure of psycho social risk assessment according to Adapted antenatal Risk Questionnaire (ANRQ) | Screening
Measure of perceived social support measured by Multidimensional Scale of Perceived Social Support (MSPSS) | 6 Months
Measure of stress using Perceived Stress Index (PSS) | 6 Months
Parenting Practices and treatment assessed by Parenting Practices and Treatment Questionnaire | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Kerker, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States